CLINICAL TRIAL: NCT05082259
Title: ASTEROID:A Phase I Trial of ASTX660 in Combination With Pembrolizumab in Patients With Solid Tumours: Utilizing Triple IAP Blockade as a Strategy to Maximize Immunogenic Cell Death and the Generation of an Efficient Adaptive Immune Response
Brief Title: ASTEROID: A Trial of ASTX660 in Combination With Pembrolizumab
Acronym: ASTEROID
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Merck Sharp & Dohme LLC (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR5199
Record Dates: First submitted 2021-10-06; First posted 2021-10-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Cancer; Cervical Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms | interventions — ASTX-660; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A-Escalation (Experimental): Increasing doses of ASTX660 in combination with a fixed dose of pembrolizumab to establish the maximum tolerated dose (MTD) of ASTX660 and Pembrolizumab when given in combination in patients with advanced solid tumours.
  escalating doses of ASTX660 will be investigated in combination with a fixed dose of Pembrolizumab (200mg). ASTX660 administration will follow a 7 day on / 14 day off pattern (ie dosing for 7 consecutive days leading up to administration of the immune check-point inhibitors). Therefore in Cycle 1, ASTX660 will be given alone from Day 1 to Day 7, followed by a 14 day break, then taken again in Cycle 2 . Each cycle will run for a period of 21 days, with ASTX660 taken always on Days 1 to 7 and Pembrolizumab given always on Day 8.
  Up to 4 dose levels of ASTX660 will be explored.
  Interventions: Drug: ASTX660; Drug: Pembrolizumab
- Part B-Expansion (Experimental): Patients in Part B will be treated at the RP2D as determined by the SRC after the initial dose escalation (Part A) has been completed. The treatment schedule will be the same as that for Part A, i.e. each cycle will be 21 days-long. Pembrolizumab will always be administered on D8 of every cycle. ASTX660 will be taken daily on Days 1-7.
  Part B will be split into 3 cohorts; Cohort B1, Cohort B2 and Cohort B3.
  Cohort B1: Patients with Immune-checkpoint refractory tumours Cohort B2: Patients with PD-L1 positive Cervical Cancer Cohort B3: Patients with Triple Negative Breast Cancer
  Interventions: Drug: ASTX660; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ASTX660 — ASTX660 will be supplied as capsules. Each hydroxylpropyl methylcellulose (HPMC) capsule contains either 30 mg or 90 mg of ASTX600 free-base equivalents, suitable for oral administration. Bottles are labelled with the capsule strength (ie, 30 mg or 90 mg) and are further distinguished by different-colored labels. Each bottle contains 14 capsules and an oxygen-absorber (not to be consumed).
  Other Names: Tolinapant
Drug: Pembrolizumab — Pembrolizumab Solution for Infusion 100 mg/vial is a liquid drug product supplied as a clear to opalescent solution, essentially free of visible particles, in Type I glass vials and manufactured using the fully formulated drug substance with L-histidine as buffering agent, polysorbate 80 as surfactant, and sucrose as stabilizer/tonicity modifier.
  Pembrolizumab Solution for Infusion can be further diluted with normal saline or 5% dextrose in the concentration range of 1 to 10 mg/mL in IV containers made of polyvinyl chloride (PVC) or non-PVC material.
  Other Names: MK-3475

SUMMARY:
This is a multi-centre Phase I dose finding and proof-of-concept study of the combination of ASTX660 together with Pembrolizumab with expansion cohorts testing preliminary efficacy in immune-refractory cancers, triple negative breast cancer (TNBC), cervical cancer, and glioblastoma.

In contrast to the existing studies combining first-generation cIAP1/2 selective Smac mimetics with immune check point inhibitors, the ASTEROID Phase I clinical trial will be the first trial utilising triple cIAP1/2 and XIAP blockade by ASTX660 as a strategy to maximise immunogenic cell death and the generation of an efficient adaptive immune response. ASTX660 is not simply being used to repeat the data already being acquired with other first generation Smac mimetics. In contrast, we will investigate more in depth the mechanisms by which ASTX660 elicits its therapeutic effects both on tumour and on the host immune system. This will be critical to determine the best strategy to pursue in future later stage tumour specific trials of IAP antagonists in combination with immunotherapy, and to ensure appropriate molecular stratification biomarkers for the greatest benefit to patients.

ELIGIBILITY:
Inclusion Criteria:

1. PART A: Patients with histologically or cytologically confirmed malignant advanced solid tumours, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient.

   PART B1: Patients with histologically or cytologically confirmed malignant advanced solid tumours (including melanoma, renal cell cancer, non-small cell lung cancer and head and neck squamous cell cancer), refractory to immune checkpoint inhibitors and for which no conventional therapy exists or is declined by the patient. Patients with other tumour types where immune checkpoint inhibitors are licensed can be considered upon discussion with the Chief Investigator.

   PART B2: Patients with histologically or cytologically confirmed cervical cancer, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient.

   PART B3: Patients with histologically or cytologically confirmed triple negative breast cancer, refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient.

   PART B4 (no longer recruiting): Patients with histologically confirmed relapsed glioblastoma (GBM). Diagnosis of GBM will be based on WHO classification of CNS tumours, 5th edition (2021):

   IDH wild type diffuse astrocytic glioma with microvascular proliferation, OR necrosis, OR one or more of the following molecular features of GBM:
   * TERT promoter mutation,
   * EGFR gene amplification,
   * 7 gain/10 loss chromosome copy number changes.

   PART B5: Patients with histologically or cytologically confirmed ER positive HER2 negative breast cancer who have progressed on CDK4/6 inhibitor therapy.

   For Immune Checkpoint inhibitor refractory tumours, participants must have progressed on treatment with an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:
   1. Has received at least 2 doses of an approved anti-PD-1/PD-L1 mAb.
   2. Has demonstrated disease progression after anti-PD-1/PD-L1 as defined by RECIST v1.1. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression (as defined in c below).
   3. Progressive disease has been documented within 24 weeks from commencing anti-PD-1/PD-L1 and no later than 12 weeks from the last dose of anti-PD-1/PD-L1 mAb.

   i) Progressive disease is determined according to iRECIST. ii) This determination is made by the investigator. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.
2. Parts A, B1, and B2: Measurable disease as assessed by imRECIST. Parts B3 and B5 : Measurable disease as assessed by imRECIST OR Evaluable disease as assessed by whole body MRI.

   Part B4: Measurable disease as assessed by RANO.
3. Patients in the ER positive HER2 negative cohort (cohort B5 ) must not have had more than two prior systemic lines of chemotherapy in the metastatic setting. There is no limitation on number of prior lines of hormonal or targeted therapies.
4. All patients with advanced solid tumours enrolled onto Part A must be willing and able to have fresh paired tissue biopsies for biomarker analysis.
5. Life expectancy of at least 12 weeks.
6. World Health Organisation (WHO) performance status of 0 or 1.
7. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) prior to the patient's first dose of IMP.

   Laboratory Test Value required Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Lymphocyte count >0.5 x 109/L Platelet count ≥ 100 x 109/L Total Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) ≤ 2.5 x (ULN) unless raised due to known metastatic liver disease in which case ≤ 5 x ULN is permissible Aspartate aminotransferase (AST) ≤ 2.5 x (ULN) unless raised due to to known metastatic liver disease in which case ≤ 5 x ULN is permissible

   Either:

   Calculated creatinine clearance

   Or:

   Creatinine

   ≥ 50 mL/min (uncorrected value)

   Or < 1.5 x upper limit of normal (ULN) Albumin >28 g/L LDH <3 x ULN Amylase ≤ ULN Lipase ≤ ULN Coagulation INR <1.5 APTT <1.5 x ULN
8. 18 years or over
9. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up
10. Female patients with reproductive potential must have a negative urine or serum pregnancy test performed within 72 hours of first dose

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy including Pembrolizumab or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) and four weeks for investigational medicinal products, except for hormonal therapy with luteinizing hormone-releasing hormone (LHRH) analogues for medical castration in patients with castrate resistant prostate cancer or ovarian suppression in pre- or peri-menopausal women with endocrine-driven breast cancer, which are permitted, and bisphosphonates or RANK ligand antagonists that are permitted for the management of bone metastases.
2. Current malignancies of other types, with the exception of adequately treated cone biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for five years or more and are deemed at negligible risk for recurrence, are eligible for the trial.
3. Ongoing Grade 2 or greater toxicities from pre-existing conditions or previous treatments. Exceptions to this are alopecia and ongoing anticoagulation therapy due to prior thromboembolic episodes.
4. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible. NB. Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
5. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] and not to donate sperm during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
6. For cohorts A, B1, B2, B3 and B5 only - Known untreated or active central nervous system (CNS) metastases (progressing or requiring corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided they meet all of the following criteria:

   * Evaluable or measurable disease outside the CNS is present.
   * Radiographic demonstration of improvement or stability upon the completion of CNS-directed therapy at least 4 weeks after completion of CNS directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the baseline disease assessment.
   * Not requiring corticosteroids.
7. For Cohort B4 only (no longer recruiting):

   * Participants with infratentorial tumors and tumors primarily located in or close to critical structures (e.g., brain stem). Patients with leptomeningeal disease.
   * Patients with evidence of raised intracranial pressure or mass effect on imaging
   * Patients unable to tolerate contrast enhanced MRI.
8. Major surgery within four weeks of the first dose of study treatment.
9. History of malabsorption syndrome or other condition that would interfere with enteral absorption.
10. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
11. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids, or current pneumonitis/interstitial lung disease.
12. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
13. Has an active autoimmune disease that has required systemic treatment in past 3 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with Sjogren's syndrome will not be excluded from the study. In addition, patients that experienced a Grade 3 or higher immune-related AE on treatment with immunotherapy will be excluded from the study. Patients that have experience a prior G2 immune-related AE on treatment will need case-by-case discussion with the CI. Patients with inactive autoimmune disease which has previously required systemic therapy, may be considered on a case-by-case basis after discussion with the sponsor.
14. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the chief Investigator. Stable use (i.e., no change in dose within 1 month prior to Day 1 of Cycle 1) of inhaled corticosteroids is allowed. Patients for cohort B4 who are on a stable dose of corticosteroids not exceeding 2mg Dexamethasone for tumour associated oedema or symptoms will be permitted to enrol on the study.
15. Has received a live vaccine within 30 days of planned start of study therapy. Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.
16. Any of the following cardiac criteria:

    1. Mean resting corrected QT interval (QTcF) > 470 msec obtained from an electrocardiogram (ECG). Known congenital QT syndrome or history of torsades de pointes.
    2. Left ventricular ejection fraction of <50% on echocardiogram.
    3. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g. complete left bundle branch block, third degree heart block. Controlled atrial fibrillation is allowed.
    4. Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association [NYHA Grade 2 or above], severe valvular disease, uncontrolled hypertension despite optimal therapy.
17. Prior bone marrow transplant or have had extensive radiotherapy to greater than 25% of bone marrow within eight weeks.
18. Participates or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study of ASTX660 and Pembrolizumab. Participation in an observational trial would be acceptable.
19. Patients with prior exposure to an IAP antagonist (Smac mimetic) will be excluded from this study. Patients with prior exposure to immunotherapy (either CTLA-4, PD-1/PD-L1 inhibitor/cellular therapy) will be permitted to enrol as long as they did not experience any immune-adverse event toxicity while on their prior immunotherapy as described in exclusion criteria 12.
20. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the Investigator's opinion.
21. Severe hypersensitivity (≥ Grade 3) to any of the IMPs and/or any of their excipients.
22. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. History of an allogenic tissue/ solid organ transplant.
24. Symptoms of COVID-19 and/or documented COVID-19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Determination of MTD and RP2D | 12 months
  To determine the Maximum Tolerated Dose (MTD) of ASTX660 in combination with Pembrolizumab based on dose-limiting toxicities (DLTs) up to 6 weeks from start of treatment and the RP2D.
Safety and tolerability | 12 months
  To determine the frequency, severity and causality of each adverse event to the combination of ASTX660 and Pembrolizumab according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Preliminary anti-tumour activity evaluation (in Part B) | 24 months
  Assessment of disease response by imRECIST criteria, clinical benefit rate, best changes in tumour size, progression-free survival and duration of response.

SECONDARY OUTCOMES:
Preliminary anti-tumour activity evaluation (in Part A) | 12 months
  Assessment of disease response by imRECIST criteria, clinical benefit rate, best changes in tumour size, progression-free survival and duration of response.
Pharmacokinetics of ASTX660 | 12 months
  Determination of the plasma levels of ASTX660 in Part A of the study, using validated assays

OTHER OUTCOMES:
Pharmacodynamics-1 | 18 months
  Determination of changes in immune cell population (using FACS) and host immune cell cytokine profile with single agent ASTX660 and the combination of ASTX660 and Pembrolizumab
Pharmacodynamics-2 | 36 months
  Determination of changes in the tumour microenvironment including changes in tumour infiltrating lymphocytes (TILs), myeloid derived suppressor cells (MDSCs) and other immune cells.
Pharmacodynamics-3 | 36 months
  Determination of changes in exploratory biomarkers including but not limited to immune transcriptome profile changes, PD-L1 expression and tumour lysate cytokine profiling in pre- and post-treatment tumour biopsies.
Pharmacodynamics-4 | 36 months
  To evaluate the effect of ASTX660 on the tumour microenvironment including the evaluation of inflammatory cytokines downstream of NF-kB in paired tumour biopsies.
Patient Reported Outcomes - Quality of Life | 36 months
  To evaluate changes in patient reported outcomes from baseline using the EORTCQLQ-C30
Overall Survival | 60 months
  To estimate the overall survival (OS) in patients receiving the combination of pembrolizumab and ASTX660.

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Lopez, MRCP, Study Director — Royal Marsden Hospital NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Cambridge University Hospitals NHS Trust, Cambridge
  - The Royal Marden NHS Foundation Trust - Drug Development Unit, Sutton
  - The Royal Marsden NHS Foundation Trust - Breast Unit, Sutton

IPD SHARING:
Plan to Share IPD: Undecided